CLINICAL TRIAL: NCT03794531
Title: Puerto Rico Observational Study of Psychosocial, Environmental, and Chronic Disease Trends
Brief Title: Psychosocial, Environmental, and Chronic Disease Trends in Puerto Rico
Acronym: PROSPECT
Status: Recruiting | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); FDI Clinical Research (Other); University of Massachusetts, Lowell (Other); San Diego State University (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Josiemer Mattei, Associate Professor of Nutrition, Harvard School of Public Health (HSPH)
Other Study IDs: 143792; R01HL143792 (NIH); R21MD013650 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2019-01-07 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Heart Diseases; Type2 Diabetes; Hypertension; Obesity; Dyslipidemias; Metabolic Syndrome; Cardiovascular Diseases; Chronic Disease; Inflammation; Psychological Stress; Physiological Stress; Depressive Symptoms; Coping Behavior; Diet Habit; Lifestyle; Food Insecurity
Keywords: Hispanics/Latinos; Minority health; Puerto Rico; Cardiovascular disease; Cardiometabolic health; Chronic disease risk factors; Disaster research; Caribbean and Latin America; Population health; Prospective study; Allostatic load; Food insecurity; Longitudinal study
MeSH Terms: conditions — Heart Diseases; Hypertension; Obesity; Dyslipidemias; Metabolic Syndrome; Cardiovascular Diseases; Chronic Disease; Inflammation; Stress, Psychological; Depression; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine, saliva, hair.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The overall goal is to identify trends and longitudinal associations in psychosocial, food-related, and cardiometabolic risk factors that can guide public health priorities and future research needs aimed at reducing cardiovascular-related disparities in Puerto Rico. To this end, investigators will establish 'PROSPECT: Puerto Rico Observational Study of Psychosocial, Environmental, and Chronic disease Trends', an island-wide, longitudinal population cohort of 2,000 adults (30-75 years) in PR recruited with a community-wide sampling strategy, and assessed in a network of several partner clinics across the island. The study will collect comprehensive data on multiple psychosocial, dietary, and food-related factors, CVD biological markers, and medical record data, with follow-up at 2-years, and will assess variations by urban-rural area and by timing before-after Maria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-75 years old at the time of enrollment
2. Non-institutionalized
3. Living in PR at the time of the first interview and the year before and not planning to move from the island within 3 years
4. Able to answer questions without assistance
5. Living in a stable dwelling

Exclusion Criteria:

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience community-wide sample of eligible adults living in all of Puerto Rico.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with self-reported medically-diagnosed chronic diseases | 4 years
  Estimate the prevalence and incidence of chronic diseases (and their dietary and psychosocial risk factors)

SECONDARY OUTCOMES:
Difference in the number of participants with self-reported medically-diagnosed chronic diseases living urban vs. rural area | 4 years
  Estimate differences in prevalence and changes in chronic diseases (and their dietary and psychosocial risk factors) in urban vs. rural area

OTHER OUTCOMES:
Risk of clinically-measured metabolic syndrome (e.g. high blood pressure, elevated adiposity, elevated blood glucose, and out-of-normal-range blood lipids), according to dietary and psychosocial risk factors | 4 years
  Determine risk of biological metabolic risk factors by changes in psychosocial factors or diet-related factors

CONTACTS AND LOCATIONS:
Locations (1):
- FDI Clinical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
IPD will be managed and distributed observing NIH and IRB policies on the dissemination and sharing of research results. Study information and requests for data will be available immediately upon the data being de-identified and properly revised for quality control on the study website.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2-years
Access Criteria: The requested data will be shared with investigators via a secured, password-protected software website.

REFERENCES:
- [Background] Mattei J, Tucker KL, Falcon LM, Rios-Bedoya CF, Kaplan RM, O'Neill HJ, Tamez M, Mendoza S, Diaz-Alvarez CB, Orozco JE, Acosta Perez E, Rodriguez-Orengo JF. Design and Implementation of the Puerto Rico Observational Study of Psychosocial, Environmental, and Chronic Disease Trends (PROSPECT). Am J Epidemiol. 2021 May 4;190(5):707-717. doi: 10.1093/aje/kwaa231. PMID 33083832
- [Background] Mattei J, Tamez M, O'Neill J, Haneuse S, Mendoza S, Orozco J, Lopez-Cepero A, Rios-Bedoya CF, Falcon LM, Tucker KL, Rodriguez-Orengo JF. Chronic Diseases and Associated Risk Factors Among Adults in Puerto Rico After Hurricane Maria. JAMA Netw Open. 2022 Jan 4;5(1):e2139986. doi: 10.1001/jamanetworkopen.2021.39986. PMID 35019984
- [Background] Lopez-Cepero A, O'Neill HJ, Marrero A, Falcon LM, Tamez M, Rodriguez-Orengo JF, Mattei J. Association between adverse experiences during Hurricane Maria and mental and emotional distress among adults in Puerto Rico. Soc Psychiatry Psychiatr Epidemiol. 2022 Dec;57(12):2423-2432. doi: 10.1007/s00127-022-02355-2. Epub 2022 Sep 1. PMID 36048184
- [Background] Xu W, Lopez-Cepero A, O'Neill HJ, Plym A, Austin SB, Mattei J. Food Insecurity Is Associated With Dysfunctional Eating Behaviors Among Adults in Puerto Rico. J Nutr Educ Behav. 2023 Sep;55(9):644-650. doi: 10.1016/j.jneb.2023.05.255. Epub 2023 Jul 1. PMID 37395692
- See also: Study website — https://www.hsph.harvard.edu/prospect/
- See also: Facebook page — https://www.facebook.com/study.prospectpr